CLINICAL TRIAL: NCT04810078
Title: A Phase 3, Open-label, Randomized, Noninferiority Trial of Subcutaneous Formulation of Nivolumab Versus Intravenous Nivolumab in Participants With Advanced or Metastatic Clear Cell Renal Cell Carcinoma Who Have Received Prior Systemic Therapy
Brief Title: A Study of Subcutaneous Nivolumab Versus Intravenous Nivolumab in Participants With Previously Treated Clear Cell Renal Cell Carcinoma That is Advanced or Has Spread
Acronym: CheckMate-67T
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA209-67T; 2020-003655-15 (EudraCT Number); U1111-1255-9514 (Registry Identifier: WHO)
Expanded Access: NCT02475382 (No longer available)
Record Dates: First submitted 2021-03-16; First posted 2021-03-22 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: BMS-936558; BMS-986298; Clear cell renal cell carcinoma; ccRCC; Nivolumab; Opdivo; rHuPH20; Subcutaneous
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (Experimental)
  Interventions: Biological: Nivolumab and rHuPH20
- Arm B (Active Comparator)
  Interventions: Biological: Nivolumab
- Arm C (Experimental)
  Interventions: Biological: Nivolumab and rHuPH20
- Arm D (Experimental)
  Interventions: Biological: Nivolumab and rHuPH20

INTERVENTIONS:
Biological: Nivolumab and rHuPH20 — Specified dose on specified days
  Other Names: BMS-986298
  Arms: Arm A; Arm C; Arm D
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Arm B

SUMMARY:
The purpose of this study is to evaluate the drug levels, efficacy, safety, and tolerability of subcutaneous nivolumab versus intravenous nivolumab in participants with previously treated clear cell renal cell carcinoma that is advanced or has spread. The purpose of this study's substudy is to evaluate drug level biocomparability of subcutaneous nivolumab manufactured using two different manufacturing processes.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histological confirmation of renal cell carcinoma (RCC) with a clear cell component, including participants who may also have sarcomatoid features
* Advanced RCC (not amenable to curative surgery or radiation therapy) or metastatic RCC (Stage IV)
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumor (RECIST) v1.1 criteria within 28 days prior to randomization
* Received no more than 2 prior systemic treatment regimens
* Intolerance or progression on or after the last treatment regimen received and within 6 months prior to randomization
* Karnofsky PS ≥ 70 at screening
* Must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Untreated, symptomatic central nervous system (CNS) metastases
* Concurrent malignancy (present during screening) requiring treatment or history of prior malignancy active within 2 years prior to randomization
* Active, known, or suspected autoimmune disease
* Known human immunodeficiency virus (HIV) positive with an acquired immunodeficiency syndrome (AIDS) defining opportunistic infection within the last year, or a current CD4 count < 350 cells/μL. Participants with HIV are eligible if:

  1. They have received established antiretroviral therapy (ART) for at least 4 weeks prior to randomization
  2. They continue on ART as clinically indicated while enrolled on study
  3. CD4 counts and viral load are monitored per standard of care by a local health care provider
  4. Inclusion of participants with HIV should be based on Investigator clinical judgment in consultation with the Medical Monitor NOTE: Testing for HIV must be performed at sites where mandated locally. HIV-positive participants must be excluded where mandated locally
* Serious or uncontrolled medical disorders including for example, active severe acute respiratory syndrome coronavirus 2 (SAR-CoV-2) infection within approximately 4 weeks prior to screening. In the case of prior SARS-CoV-2 infection, acute symptoms must have resolved based on investigator clinical judgment and, in consultation with Medical Monitor, there are no sequelae that would place the participant at a higher risk of receiving investigational treatment to be eligible
* Prior treatment with an programmed death receptor-1 (anti-PD-1), programmed death ligand-1 (anti-PD-L1), or cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways
* Treatment with any live attenuated vaccine within 30 days of first study treatment

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 681 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2027-05-10 (Estimated)

PRIMARY OUTCOMES:
Time-averaged serum concentration over 28 days (Cavgd28) | Up to 28 days
Trough serum concentration at steady-state (Cminss) | Up to 4 months

SECONDARY OUTCOMES:
Objective response rate (ORR) by Blinded Independent Central Review (BICR) with a minimum of 6 months follow-up | Up to 2 years 6 months
Trough serum concentration at day 28 (Cmind28) | At 28 days
Maximum serum concentration after the first dose (Cmax1) | Up to 7 days
Peak serum concentration at steady-state (Cmaxss) | Up to 4 months
Steady-state average serum concentration (Cavgss) | Up to 4 months
Trough concentration (Ctrough) | At week 17
Incidence of adverse events (AEs) | Up to 2 years 3 months
Incidence of serious adverse events (SAEs) | Up to 2 years 3 months
Incidence of AEs leading to discontinuation | Up to 2 years
Incidence of deaths | Up to 5 years
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to 2 years 3 months
Incidence of clinically significant changes in clinical laboratory results: Chemistry panel tests | Up to 2 years 3 months
Efficacy parameters: disease control rate (DCR) by BICR with a minimum of 6 months follow-up | Up to 2 years 6 months
Efficacy parameters: DCR by BICR with a minimum of 12 months follow-up | Up to 3 years
Efficacy parameters: DCR by BICR at end of study | Up to 5 years
Efficacy parameters: duration of response (DOR) by BICR with a minimum of 6 months follow-up | Up to 2 years 6 months
Efficacy parameters: DOR by BICR with a minimum of 12 months follow-up | Up to 3 years
Efficacy parameters: DOR by BICR at end of study | Up to 5 years
Efficacy parameters: time to objective response (TTR) by BICR with a minimum of 6 months follow-up | Up to 2 years 6 months
Efficacy parameters: TTR by BICR with a minimum of 12 months follow-up | Up to 3 years
Efficacy parameters: TTR by BICR at end of study | Up to 5 years
Efficacy parameters: progression-free survival (PFS) by BICR with a minimum of 6 months follow-up | Up to 2 years 6 months
Efficacy parameters: PFS by BICR with a minimum of 12 months follow-up | Up to 3 years
Efficacy parameters: PFS by BICR at end of study | Up to 5 years
Efficacy parameters: overall survival (OS) with a minimum of 6 months follow-up | Up to 2 years 6 months
Efficacy parameters: OS with a minimum of 12 months follow-up | Up to 3 years
Efficacy parameters: OS at end of study | Up to 5 years
Efficacy parameters: ORR by BICR with a minimum of 12 months follow-up | Up to 3 years
Efficacy parameters: ORR by BICR at end of study | Up to 5 years
Incidence of anaphylactic, hypersensitivity, and systemic infusion reactions/systemic injection reactions | Up to 2 years 3 months
Incidence of local injection- or infusion-site reactions | Up to 2 years 3 months
Percentage of participants who develop anti-nivolumab antibodies, if applicable | Up to 2 years 3 months
Percentage of participants who develop neutralizing antibodies, if applicable | Up to 2 years 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (89):
- United States (3):
  - Local Institution, Chicago, Illinois
  - Local Institution - 0025, Buffalo, New York
  - Local Institution - 0088, West Reading, Pennsylvania
- Argentina (8):
  - Local Institution - 0095, Capital Federal, Buenos Aires
  - Local Institution - 0058, Mar del Plata, Buenos Aires
  - Local Institution - 0037, Pergamino, Buenos Aires
  - Local Institution - 0079, Parana, Córdoba Province
  - Local Institution - 0030, Río Cuarto, Córdoba Province
  - Local Institution - 0066, Viedma, Río Negro Province
  - Local Institution - 0038, Buenos Aires
  - Local Institution - 0056, San Juan
- Brazil (8):
  - Local Institution - 0064, Curitiba, Paraná
  - Local Institution - 0107, Ijuí, Rio Grande do Sul
  - Local Institution - 0039, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0071, Barretos, São Paulo
  - Local Institution - 0070, São José do Rio Preto, São Paulo
  - Local Institution - 0090, Rio de Janeiro
  - Local Institution - 0081, São Paulo
  - Local Institution - 0096, São Paulo
- Chile (5):
  - Local Institution - 0084, Temuco, Región de la Araucanía
  - Local Institution - 0077, Viña del Mar, Región de Valparaíso
  - Local Institution - 0005, Santiago, Santiago Metropolitan
  - Local Institution - 0104, Santiago, Santiago Metropolitan
  - Local Institution - 0076, Santiago, Santiago Metropolitan
- Czechia (6):
  - Local Institution - 0063, Brno
  - Local Institution - 0036, Hradec Králové
  - Local Institution - 0020, Olomouc
  - Local Institution - 0099, Ostrava
  - Local Institution - 0010, Prague
  - Local Institution - 0106, Praha 8 Liben
- Local Institution - 0017, Tampere, Finland
- France (3):
  - Local Institution, Nice
  - Local Institution - 0051, Suresnes
  - Local Institution - 0068, Villejuif
- Local Institution - 0060, Tallaght, Dublin, Ireland
- Italy (11):
  - Local Institution - 0033, Cremona
  - Local Institution - 0008, Florence
  - Local Institution - 0027, Meldola
  - Local Institution - 0018, Milan
  - Local Institution, Milan
  - Local Institution - 0014, Padua
  - Local Institution - 0082, Parma
  - Local Institution - 0092, Pavia
  - Local Institution - 0100, Roma
  - Local Institution - 0091, Rome
  - Local Institution - 0057, Terni
- Mexico (7):
  - Local Institution - 0101, Torreón, Coahuila
  - Local Institution - 0089, Tlalpan, Mexico City
  - Local Institution - 0103, Monterrey, Nuevo León
  - Local Institution - 0031, Monterrey, Nuevo León
  - Local Institution - 0065, Querétaro
  - Local Institution - 0085, Querétaro
  - Local Institution - 0105, San Luis Potosí City
- New Zealand (3):
  - Local Institution - 0053, Auckland
  - Local Institution - 0041, Hamilton
  - Local Institution - 0078, Palmerston North
- Poland (7):
  - Local Institution - 0055, Biała Podlaska
  - Local Institution - 0062, Bydgoszcz
  - Local Institution - 0083, Gdansk
  - Local Institution - 0021, Krakow
  - Local Institution - 0098, Krakow
  - Local Institution - 0001, Poznan
  - Local Institution - 0023, Warsaw
- Portugal (2):
  - Local Institution - 0050, Coimbra
  - Local Institution - 0052, Lisbon
- Romania (4):
  - Local Institution - 0024, Bucharest
  - Local Institution - 0002, Cluj-Napoca
  - Local Institution - 0040, Cluj-Napoca
  - Local Institution - 0016, Craiova
- Russia (6):
  - SBIH Chelyabinsk Regional Clinical Centre of Oncology and Nuclear Medicine, Chelyabinsk
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Hertzen Moscow Oncology Research Center, Moscow
  - Local Institution, Nizghiy Novgorod
  - Budgetary Healthcare Institution of Omsk Region - Clinical Oncological Dispensary, Omsk
  - LLC Eurocityclinic, Saint Petersburg
- Spain (10):
  - Local Institution - 0048, Barcelona
  - Local Institution - 0102, Barcelona
  - Local Institution - 0049, Barcelona
  - Local Institution - 0072, Madrid
  - Local Institution - 0067, Madrid
  - Local Institution - 0074, Madrid
  - Local Institution - 0075, Madrid
  - Local Institution - 0032, Sabadell
  - Local Institution - 0086, Santander
  - Local Institution - 0059, Seville
- Turkey (Türkiye) (4):
  - Local Institution - 0035, Istanbul, Bagcilar
  - Local Institution - 0026, Ankara
  - Local Institution - 0097, Ankara
  - Local Institution - 0019, Istanbul

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04810078.html